CLINICAL TRIAL: NCT05075798
Title: A Comprehensive Retrospective Study of Cerebral MRI Anomalies in Mutated Transthyretin Amyloidosis Patients
Brief Title: Study of Cerebral MRI Anomalies in Mutated Transthyretin Amyloidosis Patients
Acronym: TTR-SNC
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2021/II-01; IRB21.09.02 (Other: IRB CHU de Nîmes)
Record Dates: First submitted 2021-09-30; First posted 2021-10-13 (Actual); Last update posted 2022-09-02 (Actual); Status verified 2022-09

CONDITIONS: Transthyretin Amyloidosis
MeSH Terms: conditions — Amyloidosis, Hereditary, Transthyretin-Related

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- group patients: Patients followed at the University Hospital of Nîmes between 2017 and 2021 for a TTR neuropathy with proven mutation, having benefited from a brain MRI.
  Interventions: Other: No intervention,

INTERVENTIONS:
Other: No intervention, — pure observational study

SUMMARY:
Transthyretin amyloidosis (aTTR) initially described as a rare disease, became the most serious hereditary polyneuropathy of adult onset and family screening has made it possible to identify and follow up many asymptomatic patients and carriers of the mutation in the TTR gene.

Considered as a systemic disease with involvement of target organs (the heart, the eye, the kidney and peripheral nervous system), it seems to be more complex for neurologists according to recent publications raising the issue of central nervous system involvement.

Indeed, TTR amyloid deposits seem to be correlated with the duration of the disease. These deposits can cause cortical damage by different mechanisms: direct TTR toxicity or as a result of pathology related to cerebral amyloid angiopathy (intraparenchymal or subarachnoid hematomas, small infarcts, hemosiderin). A small number of mutations in the TTR gene cause a rare phenotype of systemic amyloidosis, the oculoleptomeningeal form, characterized by clinical neurological symptoms: progressive dementia, epilepsy, ataxia, spastic paraparesis, stroke-like episodes.

Hypothesis of the work: the central nervous system involvement is probably underestimated on the radiological description in patients with TTR mutation.

ELIGIBILITY:
Inclusion Criteria:

* patients followed at the University Hospital of Nîmes between 2017 and 2021 for a TTR neuropathy with proven mutation, having benefited from a brain MRI.

Exclusion Criteria:

* Patients without TTR neuropathy with proven mutation, or who did not have a brain MRI.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients followed at the University Hospital of Nîmes between 2017 and 2021 for a TTR neuropathy with proven mutation, having benefited from a brain MRI.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2021-10-25 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Clinical-radiological characterization | Baseline
  Presence of signs of chronic bleeding on brain MRI (Yes/No)

CONTACTS AND LOCATIONS:
Overall Officials: Anissa MEGZARI, Study Director — Centre Hospitalier Universitaire de Nīmes
Locations (1):
- CHU de Nîmes, Nîmes, France

REFERENCES:
- [Background] Ikeda SI. [Cerebral amyloid angiopathy with familial transthyretin-derived oculoleptomeningeal amyloidosis]. Brain Nerve. 2013 Jul;65(7):831-42. Japanese. PMID 23832986
- [Result] Vieira M, Saraiva MJ. Transthyretin: a multifaceted protein. Biomol Concepts. 2014 Mar;5(1):45-54. doi: 10.1515/bmc-2013-0038. PMID 25372741
- [Result] Maia LF, Magalhaes R, Freitas J, Taipa R, Pires MM, Osorio H, Dias D, Pessegueiro H, Correia M, Coelho T. CNS involvement in V30M transthyretin amyloidosis: clinical, neuropathological and biochemical findings. J Neurol Neurosurg Psychiatry. 2015 Feb;86(2):159-67. doi: 10.1136/jnnp-2014-308107. Epub 2014 Aug 4. PMID 25091367
- [Result] Nakagawa K, Sheikh SI, Snuderl M, Frosch MP, Greenberg SM. A new Thr49Pro transthyretin gene mutation associated with leptomeningeal amyloidosis. J Neurol Sci. 2008 Sep 15;272(1-2):186-90. doi: 10.1016/j.jns.2008.05.014. Epub 2008 Jun 24. PMID 18579156
- [Result] Charidimou A, Gang Q, Werring DJ. Sporadic cerebral amyloid angiopathy revisited: recent insights into pathophysiology and clinical spectrum. J Neurol Neurosurg Psychiatry. 2012 Feb;83(2):124-37. doi: 10.1136/jnnp-2011-301308. Epub 2011 Nov 5. PMID 22056963